CLINICAL TRIAL: NCT06132646
Title: Effectiveness of a Global Proprioceptive Training After Wrist Fracture
Brief Title: Proprioceptive Training Following a Wrist Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Leire Cruz-Gambero, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RaqCan342
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Wrist Fractures; Pain
Keywords: Proprioceptive exercises; Function; Wrist fracture
MeSH Terms: conditions — Wrist Fractures; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be anonymized with a number and randomized with a web program (random.org)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients that had suffered a wrist fracture and are going to receive standard rehabilitation for the wrist.
- Experimental group (Experimental): Patients that had suffered a wrist fracture and are going to receive standard rehabilitation for the wrist.
  Interventions: Other: Proprioceptive exercises

INTERVENTIONS:
Other: Proprioceptive exercises — Specific proprioceptive exercises for the wrist that the patient has to do currently with standard rehabilitation.
  Arms: Experimental group

SUMMARY:
The goal of this randomized clinical trial is to compare how a program of proprioceptive exercises for the wrist could influence in pain, functionality and quality of life in people that have suffered a wrist fracture. The main questions it aims to answer are:

* Evaluate the effect of a specific proprioceptive program on pain and functionality.
* Study the relationship between proprioception deficit and functionality.

Intervention will be:

* Control group: participants of this group are going to receive only standard rehabilitation program after wrist fracture.
* Experimental group: participants of this group are going to receive standard rehabilitation program after distal radius fracture and a specific proprioceptive program.

Researchers will compare control and experimental group to see if a implantation of a proprioceptive program for the wrist has benefits on pain, function and quality of life.

DETAILED DESCRIPTION:
Distal radius fracture (DRF) is one of the most frequent injuries in the upper limb, corresponding to 1/6 of the total fractures of the body. It appears mostly in >50 years old women (due to osteoporosis and menopause) but it is also frequent in middle age men as a consequence of a big trauma during sport activities or working. This injury can be treated conservative of surgically, but regardless of the treatment, it always has a period of immobilization between 3 and 6 weeks.

The term "proprioception" was firstly described by Sherrington in 1906 as "perception" of body position and movement. The presence and quantity of mechanoreceptors in the joint determine its proprioceptive capacity. In the 1990s, the presence of mechanoreceptors on the wrist was described, and subsequent studies allowed us to determine that the dorsal and ulnar ligaments of the wrist have a rich innervation of mechanoreceptors. With these findings, we can hypothesize various clinical applications, both for working on wrist proprioception in the early stages of proprioceptive reeducation without risking tissue damage and for neuromuscular work after fracture consolidation, with the goal of regaining fluid and balanced movement. Previous studies on the ankle, knee, and shoulder have shown that the implementation of a proprioceptive program in the rehabilitation process can improve traumatic instability and pain. Given that the wrist shares similarities with these joints in terms of proprioceptive innervation, we can hypothesize that a specific proprioceptive exercise program for the wrist may be beneficial in the recovery after a wrist fracture.

ELIGIBILITY:
Inclusion Criteria:

* Adult (equal or more than 18 y/o).
* Suffering a wrist fracture and have passed immobilization period.
* Agree and sign informed consent.

Exclusion Criteria:

* Not had suffered a wrist fracture, being in the immobilization period or not authorized by his/her orthopedic surgeon to start with rehabilitation.
* Suffer any mental, cognitive, neurological or musculoskeletal disorder.
* Previous injury or pathology of the upper limb affected.
* Previos surgery on the upper limb affected.
* Have cervical pathology/impairment.
* Suffering from blindness.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-01-07 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in function related with daily living activities | Baseline, 4 weeks and 3 months.
  Measured with QuickDASH. 11 items, 0=no disability and 100= total disability
Change in perception of pain, referred to wrist | Baseline, 4 weeks and 3 months
  Pain measured with Numerical Rating Scale (NRS) 0= no pain and 10=worst pain
Change in hand and wrist function related with difficulties in performing daily living activities | Baseline, 4 weeks and 3 months
  Measured with Patient-rated wrist evaluation (PRWE). 15 items in 2 subscales, function (10 items) and pain (5 items). Punctuation could be from 0 to 50 in each subscale, where 50 points means worse pain/function.

SECONDARY OUTCOMES:
Change in range of motion of the wrist | Baseline, 4 weeks and 3 months.
  Active range of motion of the wrist in all planes of motion. Assessed with a goniometer.
Change in strength | Baseline, 4 weeks and 3 months.
  GRIP force. Assessed with a Jamar Dynamometer.
Change in Perception of Quality of life | Baseline, 4 weeks and 3 months
  EuroQol-5D. It has 5 dimensions, mobility, self-care, daily activities, pain and anxiety and depression. Patient determines the level of agreement with the affirmations (3 options).
Changes in proprioception, position terms | Baseline, 4 weeks and 3 months
  Measured with Joint Position Sense Test (JPST).
Changes in proprioception, strength terms | Baseline, 4 weeks and 3 months
  Measured with Force Sense Test